CLINICAL TRIAL: NCT02068586
Title: A Randomized Phase ll Study of Adjuvant Sunitinib or Valproic Acid in High-Risk Patients With Uveal Melanoma
Brief Title: Sunitinib Malate or Valproic Acid in Preventing Metastasis in Patients With High-Risk Uveal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13P.377; 2013-047 (Other: CCRRC); JT 2437 (Other: JeffTrial Number)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Ciliary Body and Choroid Melanoma, Small Size; Iris Melanoma; Stage I Intraocular Melanoma; Stage IIA Intraocular Melanoma; Stage IIB Intraocular Melanoma; Stage IIIA Intraocular Melanoma; Stage IIIB Intraocular Melanoma; Stage IIIC Intraocular Melanoma; Stage I Uveal Melanoma AJCC V7; Stage II Uveal Melanoma AJCC V7; Stage III Uveal Melanoma AJCC V7
MeSH Terms: conditions — Uveal Melanoma | interventions — Sunitinib; Valproic Acid; Epilim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sunitinib- (Cohort 1, Arm I) (Experimental): Patients receive sunitinib malate PO daily for 6 months in the absence of disease progression or unacceptable toxicity
  Quality-of-Life Assessment-Ancillary studies
  - Laboratory Biomarker Analysis-Correlative studies
  Interventions: Drug: Sunitinib
- Valproic acid- (Cohort 1, Arm II) (Experimental): Patients receive valproic acid PO daily for 6 months in the absence of disease progression or unacceptable toxicity
  Quality-of-Life Assessment-Ancillary studies
  Laboratory Biomarker Analysis-Correlative studies
  Interventions: Drug: Valproic Acid
- Sunitinib Malate (Cohort 2) (Experimental): Patients receive sunitinib malate PO daily for 12 months in the absence of disease progression or unacceptable toxicity
  Quality-of-Life Assessment-Ancillary studies
  Laboratory Biomarker Analysis-Correlative studies
  Interventions: Drug: Sunitinib Malate
- Sunitinib Malate + Valproic Acid (Cohort 3) (Active Comparator): Patients receive sunitinib malate PO daily and valproic acid PO daily for 12 months in the absence of disease progression or unacceptable toxicity.
  Quality-of-Life Assessment-Ancillary studies
  Laboratory Biomarker Analysis-Correlative studies
  Interventions: Drug: Sunitinib Malate + Valproic Acid

INTERVENTIONS:
Drug: Sunitinib — Given PO
  Other Names: Sunitinib malate; Sutent; SU11248; 341031-54-7 Butanedioic acid
  Arms: Sunitinib- (Cohort 1, Arm I)
Drug: Valproic Acid — Given PO
  Other Names: VPA; Valproate; Valproate sodium; Depakote; Epilim; Valparin; Valpro; Stavzor; Depakene; Di-n-propylacetic Acid
  Arms: Valproic acid- (Cohort 1, Arm II)
Drug: Sunitinib Malate — Given PO
  Other Names: sunitinib; Sutent; SU011248
  Arms: Sunitinib Malate (Cohort 2)
Drug: Sunitinib Malate + Valproic Acid — Given PO
  Other Names: Sunitinib Malate; sunitinib; Sutent; SU011248; Valproic Acid; VPA; Valproate; Valproate sodium; Depakote; Epilim; Valparin; Valpro; Stavzor; Depakene; Di-n-propylacetic Acid
  Arms: Sunitinib Malate + Valproic Acid (Cohort 3)

SUMMARY:
This randomized phase II trial studies how well sunitinib malate or valproic acid works in preventing high-risk uveal (eye) melanoma from spreading to other parts of the body. Sunitinib malate may stop the transmission of growth signals into tumor cells and prevents these cells from growing. Valproic acid may change the expression of some genes in uveal melanoma and suppress tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of adjuvant sunitinib malatate (sunitinib) and adjuvant valproic acid used for 6 months to improve overall survival (OS) at 2 years in patients with high risk uveal melanoma. (Cohort 1) II. To assess the efficacy of adjuvant sunitinib used for 12 months to improve 1.5-year relapse free survival (RFS) in patients with high-risk uveal melanoma. (Cohort 2) III. To assess whether the combination of sunitinib and valproic acid used for 12 months improve the 2-year relapse free survival (RFS) in patients with high-risk uveal melanoma. (Cohort 3)

SECONDARY OBJECTIVES:

I. To assess the efficacy of adjuvant sunitinib, in terms of RFS and adjuvant valproic acid used for 6 months in preventing the development of distal metastases in patients with high risk uveal melanoma. (Cohort 1) II. To assess the efficacy of adjuvant sunitinib, in terms of OS, used for 12 months in patients with high risk uveal melanoma. (Cohort 2) III. To assess the efficacy of adjuvant sunitinib in combination with valproic acid, in terms of OS in patients with high risk uveal melanoma. (Cohort 3) IV. To confirm the safety and tolerability of 6 months of adjuvant sunitinib and adjuvant valproic acid. (Cohort 1) V. To confirm the safety and tolerability of 12 months of adjuvant sunitinib. (Cohort 2) VI. To confirm the safety and tolerability of 12 months of adjuvant sunitinib and valproic acid. (Cohort 3)

TERTIARY OBJECTIVES:

I. To determine whether blood myeloid-derived suppressor cells (MDSCs) concentration and other inflammatory cytokines correlates with OS and RFS.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: Participants are randomized to 1 of 2 arms.

ARM I: Patients receive sunitinib malate orally (PO) daily for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive valproic acid PO daily for 6 months in the absence of disease progression or unacceptable toxicity.

COHORT 2: Patients receive sunitinib malate PO daily for 12 months in the absence of disease progression or unacceptable toxicity.

COHORT 3: Patients receive sunitinib malate PO daily and valproic acid PO daily for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Histologically-confirmed primary uveal melanoma
* Definitive local treatment for primary tumor, including surgical resection (enucleation) or radiation therapy (radioactive plaque or external proton beam)
* High risk for distal recurrence defined as any of the following conditions: A) Confirmed both monosomy 3 and 8q amplification; B) Class II tumor
* Less than 6 months from the date that local treatment (surgical or radiation) of the primary tumor was finalized
* Karnofsky performance status (PS) scores of 70 or greater
* If female, no pregnancy
* If of child-bearing potential (< one year post-menopausal), must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, condom, diaphragm with spermicidal, cervical cap, abstinence or sterile sex partner) from the time informed consent is signed (women only) or the time of initiation of sunitinib (sunitinib malate) (men only); both men and women must agree to continue using such precautions while receiving sunitinib or valproic acid and for 30 days after the final dose
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 8 g/dl
* Serum creatinine < 1.5 times upper limit of normal range (ULN) or creatinine clearance >= 40 ml/min
* Serum bilirubin < 1.5 times ULN
* Serum albumin > 2.0 g/dl
* Adequate cardiac function (ejection fraction [EF] > 50%) based on multi gated acquisition (MUGA) scan or 2 dimensional-echocardiogram (2D-Echo)
* Life expectancy of at least 5 years

Exclusion Criteria:

* Other malignancy within 5 years, except curatively treated non-melanomatous skin cancer, curatively treated carcinoma in situ of the uterine cervix, or early stage (stage I or IIa) prostate cancer
* Metastatic uveal melanoma
* History of severe allergic reaction to sunitinib or valproic acid; inability to receive sunitinib or valproic acid
* Previous treatment with sunitinib or valproic acid for uveal melanoma
* Active treatment with valproic acid for non-oncological conditions, if this cannot be safely switched to an alternative agent
* Active epilepsy or convulsive conditions that require continuous use of anticonvulsants
* Patients with known urea cycle disorders (i.e.: ornithine transcarbamylase deficiency)
* Severe cardiovascular disease within 6 months, including myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebro-vascular accident or transient ischemic attack, pulmonary embolism, life threatening arrhythmias, uncontrollable hypertension or QT prolongation syndrome
* Active liver disease (i.e., cirrhosis, viral or autoimmune hepatitis, etc.)
* Pregnancy or unwillingness to stop breast-feeding
* Prior myelosuppressive chemotherapy or other investigational drug therapy within the last 6 months prior to initiation of sunitinib or valproic acid
* Current evidence of hematemesis, melena or gross hematuria
* History or presence of any significant bleeding disorders
* Concurrent use of a strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitor or inducer; these medications should be discontinued or switched to a different medication with a weaker CYP3A4 interaction prior to enrollment into the study; if patients need to continue the same medication(s), they are excluded from the study
* Chronic usage of aspirin greater than 81 mg/day
* Unable to render informed consent and to follow protocol requirements
* Any other medical condition(s) that, at the discretion of the principal investigator (PI), would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (Cohort 1) | Time of definitive treatment of the primary tumor until death from any cause, assessed at 2 years
  OS distribution will be summarized using the method of Kaplan-Meier and the 2-year OS rate with two-sided 90% confidence interval (CI) will be provided. OS will be compared to the historic OS using a one-sample log-rank test.
Relapse-free survival (RFS) (Cohort 2 and 3) | Time of definitive treatment of the primary tumor until confirmed metastatic relapse or death from any cause, assessed at 2 years
  RFS distribution will be summarized using the method of Kaplan-Meier. 1.5-year, 2-year PFS rate will be computed with the corresponding two-sided 90% confidence intervals. OS and RFS will be compared to the null hypothesis OS or RFS using a one-sided one-sample Brookmeyer-Crowley test with alpha 0.05

SECONDARY OUTCOMES:
Relapse-free survival (Cohort 1) | Time of definitive treatment of the primary tumor until confirmed metastatic relapse or death from any cause, assessed at 2 years
  RFS distribution will be summarized using the method of Kaplan-Meier, and two-sided 90% confidence interval (CI) will be provided.
Overall survival (Cohort 2) | Time of definitive treatment of the primary tumor until death from any cause, assessed at 2 years
  OS distribution will be summarized using the method of Kaplan-Meier and the 2-year OS rate with two-sided 90% confidence interval (CI) will be provided. OS will be compared to the historic OS using a one-sample log-rank test.
Tolerability, defined as the proportion of patients able to complete 6 months of treatment, including those who underwent dose reduction | 6 months
  Proportion of patients completing six months of treatment will be summarized using descriptive statistics.
Incidence of toxicity assessed according to the National Institute of Health Common Terminology Criteria for Adverse Events (NIH CTCAE) version 4.0 | Up to 5 years
  Type and grade of toxicity will be assessed on every schedule visit and recorded based on NIH CTCAE 4.0 grading system. Descriptive statistics will be used to summarized type and grade of toxicity.
Quality of life (QOL) assessed by Functional Assessment of Cancer Therapy-General (FACT-G) questionnaires | Up to 6 months
  The FACT-G questionnaires will be scored at baseline, 1 month, 3 months, and 6 months. The difference between two treatment groups will be analyzed with standard t-test at individual evaluation points. Average QOL scores during the study will be calculated and compared between the treatment groups. To estimate the magnitude of the difference between treatment groups, the standardized effect size and minimally important difference will be used. Repeated-measures mixed-effects models with random intercepts and slopes will be used to assess treatment differences in QOL measures over time.

CONTACTS AND LOCATIONS:
Overall Officials: Takami Sato, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org